CLINICAL TRIAL: NCT01868685
Title: An Exploratory, Randomized, Double-blind, Placebo-controlled Study to Investigate the Effect of BYM338 on Muscle in Patients Requiring Prolonged Mechanical Ventilation
Brief Title: Study of Muscle Effects of BYM338 in Mechanically Ventilated Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CBYM338X2207
Record Dates: First submitted 2013-04-12; First posted 2013-06-04 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Mechanical Ventilation
Keywords: Muscle, anabolism, cachexia, respiratory failure, diaphragm
MeSH Terms: conditions — Cachexia; Respiratory Insufficiency | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BYM338 (Experimental)
  Interventions: Drug: BYM338

INTERVENTIONS:
Drug: BYM338 — BYM338
  Arms: BYM338
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of BYM338 on muscle mass and function in Group III failure to wean patients, as compared to placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* Adults on mechanical ventilation for at least 7 days with a tracheostomy in place for >24 hours.
* Expected to survive at least 14 days.
* Receiving adequate nutritional support, defined as at least 20 kcal/kg and 0.6 g/kg protein per day (unless lower protein intake required by clinical status).

Exclusion Criteria:

* Patients deemed to be terminal wean patients.
* Patients who have progressive neuromuscular degenerative disorders.
* Patients who are comatose.
* Evidence of unstable medical status.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in thigh muscle thickness | After 14 days

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | After 12 weeks
Sparse sampling of BYM338 serum levels to assess pharmacokinetic profile in mechanically ventilated patients | After 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals